CLINICAL TRIAL: NCT04782375
Title: A Multicenter Prospective Open-label Single Arm Trial to Safely Discontinue Antiviral Treatment in Patients With Chronic Hepatitis B With a Comparison to Matched Historical Controls (ADAPT)
Brief Title: Safely Discontinue Antiviral Treatment in Patients With Chronic Hepatitis B
Acronym: ADAPT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Suk Lim, PhD, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AMC 2021-0135
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-12

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm A (Experimental): discontinue antiviral treatment
  Interventions: Drug: Stop group

INTERVENTIONS:
Drug: Stop group — discontinue antiviral treatment
  Other Names: discontinue antiviral treatment

SUMMARY:
Multicenter, Prospective Open-label Single Arm Trial Chronic hepatitis B male and female adults on antiviral treatment for hepatitis B, without cirrhosis who are currently HBV DNA (-) and HBeAg (-) To evaluate the safety and efficacy of stopping long-term antiviral therapy in chronic hepatitis B patients without cirrhosis who are currently HBV DNA (-) and HBeAg (-)

DETAILED DESCRIPTION:
This clinical trial is a multicenter, Prospective Open-label Single Arm Trial to compare the short-term clinical outcome between stopping and continuing antiviral treatment in chronic hepatitis B patients without cirrhosis who are currently HBV DNA (-) and HBeAg (-) Approximately 140 subjects meeting eligibility criteria will be enrolled a Intervention Arm as below;

* Intervention Arm: 140 subjects, discontinue antiviral treatment (stop group)
* Historical cohort: 700 subjects, continue antiviral treatment

Stop group is scheduled to be followed up to 12months. Patients in the stop group were retreated with nucleos(t)ide analogues that had been prescribed previously if they fulfill one of the following criteria: 1) HBV DNA >2,000 IU/mL, 2) progression to liver cirrhosis, or 3) development of hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to study entry
2. Age ≥19 years and ≤65 years at the time of screening
3. HBsAg titer <3,000 IU/mL at the time of screening
4. Antiviral treatment continued at least 2 years and HBeAg (-) at the time of screening
5. Undetectable HBV DNA level at the time of screening
6. Serum ALT level <80 IU/mL at the time of screening
7. Estimated creatinine clearance ≥30 ml/min (by calculation of creatinine clearance or using the CKD-EPI equation)
8. Ability to comply with all study requirements

Exclusion Criteria:

1. Confirmed known co-infection with HCV, HIV, or HDV
2. Evidence of liver cirrhosis defined as meeting any of the following criteria:
3. Current alcohol (60g/day) or substance abuse judged by the investigator that will potentially interfere with subject compliance (1) Splenomegaly (>12 cm) assessed by ultrasound, CT, or MRI (2) Fibroscan ≥9.0 kPa (3) Platelet count <150,000/mm3 However, if the above criteria were satisfied at the time of antiviral treatment initiation, subjects may be eligible if they have low possibility of having liver cirrhosis with improvement in liver function by long-term antiviral treatment, following the opinion of the investigator.
4. Any history of clinical hepatic decompensation (e.g., ascites, encephalopathy, variceal hemorrhage) within 12 months prior to the screening or Child-Pugh score of ≥7 at the time of screening
5. Currently on or have received therapy with Interferon or immunosuppressant (including systemic chemotherapy) within 12 months prior to the screening
6. Requirement for chronic use of systemic immunosuppressant including, but not limited to, corticosteroid (prednisone equivalent of >40 mg/day for >2 weeks), azathioprine, or monoclonal antibodies
7. Received solid organ or bone marrow transplant
8. Any other clinical conditions (cardiovascular, respiratory, neurologic, or renal conditions) or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements.
9. History or current evidence of hepatocellular carcinoma (HCC), or high α-fetoprotein (AFP) > 20 ng/mL. (But, the patients with AFP > 20 ng/mL can be enrolled and there is no evidence of HCC by dynamic CT or MRI perfomred within 4 months prior to the screening)
10. Malignancy other than hepatocellular carcinoma within the 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (within 2 years prior to screening with confirmation of no evidence of disease). Subjects under evaluation for possible malignancy are not eligible.
11. Concurrent enrollment in another clinical study for other type of antiviral treatment for CHB or immune modulatory drug within 3 months prior to Screening, participation to an observational (non-interventional) clinical studies or interventional studies not using anti-HBV or immune modulatory drugs, or during the follow-up period of an interventional study are not exclusion criteria.
12. Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
virological relapse | Change from baseline in HBV DNA result at 6month and 12month
  Proportion of virological relapse defined as HBV DNA ≥2,000 IU/mL

SECONDARY OUTCOMES:
hospital admission | From baseline, clinical events will be collected within 12month
  Proportion of liver-related unexpected hospital admission
Proportion of clinical relapse | at 6month and 12 month
  Proportion of clinical relapse (HBV DNA ≥2,000 IU/mL and ALT ≥80 IU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Suk Lim, PhD, Principal Investigator — Asan Medical Center
Locations (9):
- South Korea (9):
  - Kyungpook National University Hospital, Daegu
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung-Hee University Hospital, Seoul
  - Samsung Medical center, Seoul
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No